CLINICAL TRIAL: NCT05720169
Title: Fetal, Obstetrics and Reproduction Genomics
Acronym: FORgenomics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundación Ginemed (Other)
Collaborators: Hospitales Universitarios Virgen del Rocío (Other); University of Seville (Other); Clínicas Ginemed (Unknown); FIRST - Fetal, IVF and Reproduction Simulation Training Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0001
Record Dates: First submitted 2023-01-29; First posted 2023-02-09 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Preeclampsia; Intrauterine Growth Restriction; Placental Disease
Keywords: Preeclampsia; Intrauterine Growth Restriction; Genomics
MeSH Terms: conditions — Pre-Eclampsia; Fetal Growth Retardation; Placenta Diseases | interventions — Ultrasonography, Doppler; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Doppler ultrasound — Doppler ultrasound at 13, 16, 20 and 26 weeks for assessment of uterine arteries according to ISUOG criteria.
Diagnostic Test: Blood sample — Blood sampling at 13, 16, 20, 26 weeks of gestation to determine the sFlt-1/PlGF ratio
Diagnostic Test: Blood sample — Blood sampling at week 13 for DNA extraction for genomic studies
Diagnostic Test: Doppler ultrasound — Fetal morphological ultrasound at 13, 16 and 20 weeks.

SUMMARY:
The purpose of this study is to determine the impact of a clinical screening strategy and genomic analysis of the factors involved in Placental Dysfunction (Preeclampsia and IUGR) in women of advanced maternal age undergoing assisted reproduction techniques (ART), specifically, in vitro fertilization (IVF) and oocyte donation.

DETAILED DESCRIPTION:
Given society's shift towards later childbearing, partly related to increased career development, women are increasingly delaying childbearing and, as a result, face declining biological fertility and increased maternal morbidity and adverse perinatal pregnancy outcomes, as well as increased use of ART. Preeclampsia (PE) complicates 2% of pregnancies and is a leading cause of severe maternal and perinatal complications. There is no curative treatment, and the only recognized beneficial primary prevention is low-dose aspirin. Finding an effective method of predicting and preventing placental dysfunction (PD) in women of advanced maternal age undergoing ART remains a challenge.

The investigators believe that maternal and perinatal complications in this group of pregnant women could be detected preclinically and allow early preventive actions.

On the other hand, establishing a differentiated genomic pattern in this group of patients would allow preventive actions both pregestational and during gestation. Furthermore, FORgenomics can be used to externally validate a prediction model for the development of PE and IUGR in pregnancy after IVF/ovodon. Our results could be applicable in most healthcare settings and have important implications for maternal-fetal health.

The justification and hypothesis of this proposal is: (1) maternal and perinatal complications in this group of pregnant women could be detected preclinically and allow preventive actions by systematic screening based on Doppler ultrasound of uterine arteries and anti-angiogenic factors (sFlt-1/PlGF ratio) at 13, 16, 20 and 26 weeks to identify pregnant women at high risk for developing PE; (2) morphological ultrasound at 13, 16 and 20 weeks would help to establish a standardized procedure for early detection of congenital anomalies and (3) establishing a differentiated genomic pattern in this group of patients would allow preventive actions both pregestational and during gestation.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Age ≥40 years
* Signed informed consent
* Gestation obtained by IVF or ovodonation

Exclusion Criteria:

* Non-ongoing pregnancy
* Gestation obtained by artificial insemination
* Naturally obtained gestation, without ART
* Multiple pregnancy
* Pregnancies complicated by major fetal abnormality identified at the first-trimester ultrasound
* Age <18 years
* Poor understanding of the Spanish or English languages
* Refusal in informed consent to participate in the study
* Participation in another intervention study that could modify follow-up

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sample
  1. Virgen del Rocío Hospital Area: according to the data obtained from the pregnant women who start the pregnancy process in the Andalusian Congenital Anomalies Screening Program (PACAC) in 2021, we expect a total population of 165 pregnant women per year with age at the start of pregnancy equal to or greater than 40 years, and whose pregnancy was obtained through IVF or ovodonation.
  2. Clínicas Ginemed: according to the data obtained from the report of Ginemed Clinics for the year 2021, we expect a total population of 150 pregnant women per year with an age at the onset of pregnancy equal to or greater than 40 years old, and whose gestation was obtained through IVF or ovodonation.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with preeclampsia (PE) during pregnancy | ≥20 weeks to <37 weeks of gestation
  Defined as systolic blood pressure ≥ 140mmHg or diastolic blood pressure ≥ 90mmHg with an interval of at least 4 h after 20 weeks' gestation plus any of the following: (i) proteinuria (>300 mg/24 h) or a urine protein/creatinine ratio > 0.3 mg/mmol); (ii) end-organ dysfunction: systolic blood pressure > 160 mmHg, diastolic blood pressure >110 mmHg, platelet count <100x109/L, blood alanine and aspartate transaminases >70 IU/L, serum creatinine >1. 1 mg/dL, lactate dehydrogenase >700 IU/L, right upper quadrant or epigastric pain, dyspnea and/or cerebral/visual disturbances. Or (iii) utero-placental dysfunction (estimated fetal weight <3rd centile or <10th centile with abnormal uterine or umbilical Doppler [pulsatility index >95th centile]) as defined by the International Society for the Study of Hypertension in Pregnancy (ISSHP) with minor adaptations for study purposes.
Number of fetuses diagnosed with intrauterine growth restriction (IUGR) during pregnancy | ≥20 weeks to <37 weeks of gestation
  IUGR will be defined by the following criteria: Estimated fetal weight (EFW) between percentile (p) 3 and p 10 with Doppler alteration (uterine arteries > p 95 or cerebroplacental index < p 5, or middle cerebral artery < p 5, or umbilical artery > p 95). PFE < p 3 independently of feto-maternal Doppler.

SECONDARY OUTCOMES:
Number of fetuses and newborns with severe perinatal morbidity | From birth up to 7 days of life
  Defined by a composite including any of the following: premature placental abruption, severe fetal growth restriction (birth weight <3rd centile), perinatal mortality, an Apgar score at 5'< 7.0, arterial pH less than 7.10, need for respiratory support within 72 hours of birth, neonatal intraventricular hemorrhage grade III/IV, necrotizing, periventricular leukomalacia, sepsis, bronchopulmonary dysplasia or encephalopathy due to hypoxic ischemic enterocolitis. Days of admission to ICU.
Cesarean section rate | During birth
  Type of delivery and cesarean section rate will be recorded.
Number of Participants with pregnancy-related maternal morbidity | From conception up to 4 days after birth
  defined by a composite including any of the following: (i) HELLP syndrome (lactate dehydrogenase [LDH] >700 IU/L, AST at twice normal values, and platelet count <100x109/L); (ii) central nervous system dysfunction (eclampsia, Glasgow Coma Score <13, stroke, reversible ischemic neurologic deficit, or cortical blindness); (iii) hepatic dysfunction (INR >1. 2 in the absence of disseminated intravascular coagulation, MELD score >10, or hepatic hematoma or rupture); (iv) renal dysfunction (dialysis, serum creatinine concentration greater than 150 μmol/L, or diuresis <0.5 mL/kg/h for 12 hours, according to renal failure by RIFLE criteria; or need for furosemide treatment to maintain diuresis >0. 5 mL/kg/h for 3 hours); (v) respiratory dysfunction (pulmonary edema, need for invasive or noninvasive mechanical ventilation, need for oxygen concentration greater than 50% for more than 1 hour, or severe respiratory distress [without pulmonary edema criteria but with presence of dyspnea,
Maternal experience and psychological impact | From conception up to 4 days after birth
  It will be assessed by:
  - WHO Five Well-Being Index (WHO), Spanish version of 1998, applied at week 26. A brief self-assessment questionnaire on a person's perception of well-being over a specific period of time.
Maternal anxiety and psychological impact | From conception up to 4 days after birth
  It will be assessed by:
  - Spielberger State-Trait Anxiety Questionnaire (STAI), in its Spanish adaptation applied in the 26th week of gestation. One of the first instruments validated in Spain and one of the most widely used by many researchers, it comprises two differentiated self-assessment scales: State Anxiety (SA), referring to a transitory anxious state that a person may feel in specific situations; and Trait Anxiety (RA), which characterizes a more or less stable anxious tendency that distinguishes people in their tendency to perceive situations as threatening.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Usta IM, Nassar AH. Advanced maternal age. Part I: obstetric complications. Am J Perinatol. 2008 Sep;25(8):521-34. doi: 10.1055/s-0028-1085620. Epub 2008 Sep 4. PMID 18773378
- [Background] Zegers-Hochschild F, Adamson GD, de Mouzon J, Ishihara O, Mansour R, Nygren K, Sullivan E, Vanderpoel S; International Committee for Monitoring Assisted Reproductive Technology; World Health Organization. International Committee for Monitoring Assisted Reproductive Technology (ICMART) and the World Health Organization (WHO) revised glossary of ART terminology, 2009. Fertil Steril. 2009 Nov;92(5):1520-4. doi: 10.1016/j.fertnstert.2009.09.009. Epub 2009 Oct 14. PMID 19828144
- [Background] Thoma ME, McLain AC, Louis JF, King RB, Trumble AC, Sundaram R, Buck Louis GM. Prevalence of infertility in the United States as estimated by the current duration approach and a traditional constructed approach. Fertil Steril. 2013 Apr;99(5):1324-1331.e1. doi: 10.1016/j.fertnstert.2012.11.037. Epub 2013 Jan 3. PMID 23290741
- [Background] Cedars MI, Taymans SE, DePaolo LV, Warner L, Moss SB, Eisenberg ML. The sixth vital sign: what reproduction tells us about overall health. Proceedings from a NICHD/CDC workshop. Hum Reprod Open. 2017 Jul 12;2017(2):hox008. doi: 10.1093/hropen/hox008. eCollection 2017. PMID 30895226
- [Background] American College of Obstetricians and Gynecologists' Committee on Obstetric Practice; Committee on Genetics; U.S. Food and Drug Administration. Committee Opinion No 671: Perinatal Risks Associated With Assisted Reproductive Technology. Obstet Gynecol. 2016 Sep;128(3):e61-8. doi: 10.1097/AOG.0000000000001643. PMID 27548556
- [Background] Pandey S, Shetty A, Hamilton M, Bhattacharya S, Maheshwari A. Obstetric and perinatal outcomes in singleton pregnancies resulting from IVF/ICSI: a systematic review and meta-analysis. Hum Reprod Update. 2012 Sep-Oct;18(5):485-503. doi: 10.1093/humupd/dms018. Epub 2012 May 19. PMID 22611174
- [Background] Schieve LA, Cohen B, Nannini A, Ferre C, Reynolds MA, Zhang Z, Jeng G, Macaluso M, Wright VC; Massachusetts Consortium for Assisted Reproductive Technology Epidemiologic Research (MCARTER). A population-based study of maternal and perinatal outcomes associated with assisted reproductive technology in Massachusetts. Matern Child Health J. 2007 Nov;11(6):517-25. doi: 10.1007/s10995-007-0202-7. Epub 2007 Mar 8. PMID 17345154
- [Background] Qin JB, Sheng XQ, Wang H, Chen GC, Yang J, Yu H, Yang TB. Worldwide prevalence of adverse pregnancy outcomes associated with in vitro fertilization/intracytoplasmic sperm injection among multiple births: a systematic review and meta-analysis based on cohort studies. Arch Gynecol Obstet. 2017 Mar;295(3):577-597. doi: 10.1007/s00404-017-4291-2. Epub 2017 Feb 6. PMID 28168654
- [Background] Helmerhorst FM, Perquin DA, Donker D, Keirse MJ. Perinatal outcome of singletons and twins after assisted conception: a systematic review of controlled studies. BMJ. 2004 Jan 31;328(7434):261. doi: 10.1136/bmj.37957.560278.EE. Epub 2004 Jan 23. PMID 14742347
- [Background] Jackson RA, Gibson KA, Wu YW, Croughan MS. Perinatal outcomes in singletons following in vitro fertilization: a meta-analysis. Obstet Gynecol. 2004 Mar;103(3):551-63. doi: 10.1097/01.AOG.0000114989.84822.51. PMID 14990421
- [Background] McDonald SD, Han Z, Mulla S, Murphy KE, Beyene J, Ohlsson A; Knowledge Synthesis Group. Preterm birth and low birth weight among in vitro fertilization singletons: a systematic review and meta-analyses. Eur J Obstet Gynecol Reprod Biol. 2009 Oct;146(2):138-48. doi: 10.1016/j.ejogrb.2009.05.035. Epub 2009 Jul 4. PMID 19577836
- [Background] Qin J, Liu X, Sheng X, Wang H, Gao S. Assisted reproductive technology and the risk of pregnancy-related complications and adverse pregnancy outcomes in singleton pregnancies: a meta-analysis of cohort studies. Fertil Steril. 2016 Jan;105(1):73-85.e1-6. doi: 10.1016/j.fertnstert.2015.09.007. Epub 2015 Oct 9. PMID 26453266
- [Background] Kawwass JF, Monsour M, Crawford S, Kissin DM, Session DR, Kulkarni AD, Jamieson DJ; National ART Surveillance System (NASS) Group. Trends and outcomes for donor oocyte cycles in the United States, 2000-2010. JAMA. 2013 Dec 11;310(22):2426-34. doi: 10.1001/jama.2013.280924. PMID 24135860
- [Background] Jeve YB, Potdar N, Opoku A, Khare M. Donor oocyte conception and pregnancy complications: a systematic review and meta-analysis. BJOG. 2016 Aug;123(9):1471-80. doi: 10.1111/1471-0528.13910. Epub 2016 Feb 8. PMID 26854328
- [Background] Jacobsson B, Ladfors L, Milsom I. Advanced maternal age and adverse perinatal outcome. Obstet Gynecol. 2004 Oct;104(4):727-33. doi: 10.1097/01.AOG.0000140682.63746.be. PMID 15458893
- [Background] Kenny LC, Lavender T, McNamee R, O'Neill SM, Mills T, Khashan AS. Advanced maternal age and adverse pregnancy outcome: evidence from a large contemporary cohort. PLoS One. 2013;8(2):e56583. doi: 10.1371/journal.pone.0056583. Epub 2013 Feb 20. PMID 23437176
- [Background] Yogev Y, Melamed N, Bardin R, Tenenbaum-Gavish K, Ben-Shitrit G, Ben-Haroush A. Pregnancy outcome at extremely advanced maternal age. Am J Obstet Gynecol. 2010 Dec;203(6):558.e1-7. doi: 10.1016/j.ajog.2010.07.039. Epub 2010 Oct 20. PMID 20965486
- [Background] Reddy UM, Ko CW, Willinger M. Maternal age and the risk of stillbirth throughout pregnancy in the United States. Am J Obstet Gynecol. 2006 Sep;195(3):764-70. doi: 10.1016/j.ajog.2006.06.019. PMID 16949411
- [Background] Lean SC, Derricott H, Jones RL, Heazell AEP. Advanced maternal age and adverse pregnancy outcomes: A systematic review and meta-analysis. PLoS One. 2017 Oct 17;12(10):e0186287. doi: 10.1371/journal.pone.0186287. eCollection 2017. PMID 29040334
- [Background] Wennberg AL, Opdahl S, Bergh C, Aaris Henningsen AK, Gissler M, Romundstad LB, Pinborg A, Tiitinen A, Skjaerven R, Wennerholm UB. Effect of maternal age on maternal and neonatal outcomes after assisted reproductive technology. Fertil Steril. 2016 Oct;106(5):1142-1149.e14. doi: 10.1016/j.fertnstert.2016.06.021. Epub 2016 Jul 9. PMID 27399261
- [Background] Wen J, Jiang J, Ding C, Dai J, Liu Y, Xia Y, Liu J, Hu Z. Birth defects in children conceived by in vitro fertilization and intracytoplasmic sperm injection: a meta-analysis. Fertil Steril. 2012 Jun;97(6):1331-7.e1-4. doi: 10.1016/j.fertnstert.2012.02.053. Epub 2012 Apr 3. PMID 22480819
- [Background] Boulet SL, Kirby RS, Reefhuis J, Zhang Y, Sunderam S, Cohen B, Bernson D, Copeland G, Bailey MA, Jamieson DJ, Kissin DM; States Monitoring Assisted Reproductive Technology (SMART) Collaborative. Assisted Reproductive Technology and Birth Defects Among Liveborn Infants in Florida, Massachusetts, and Michigan, 2000-2010. JAMA Pediatr. 2016 Jun 6;170(6):e154934. doi: 10.1001/jamapediatrics.2015.4934. Epub 2016 Jun 6. PMID 27043648
- [Background] Giorgione V, Parazzini F, Fesslova V, Cipriani S, Candiani M, Inversetti A, Sigismondi C, Tiberio F, Cavoretto P. Congenital heart defects in IVF/ICSI pregnancy: systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2018 Jan;51(1):33-42. doi: 10.1002/uog.18932. PMID 29164811
- [Background] Society for Maternal-Fetal Medicine (SMFM). Electronic address: pubs@smfm.org; Martins JG, Biggio JR, Abuhamad A. Society for Maternal-Fetal Medicine Consult Series #52: Diagnosis and management of fetal growth restriction: (Replaces Clinical Guideline Number 3, April 2012). Am J Obstet Gynecol. 2020 Oct;223(4):B2-B17. doi: 10.1016/j.ajog.2020.05.010. Epub 2020 May 12. PMID 32407785
- [Background] Gordijn SJ, Beune IM, Thilaganathan B, Papageorghiou A, Baschat AA, Baker PN, Silver RM, Wynia K, Ganzevoort W. Consensus definition of fetal growth restriction: a Delphi procedure. Ultrasound Obstet Gynecol. 2016 Sep;48(3):333-9. doi: 10.1002/uog.15884. PMID 26909664
- [Background] Cantwell R, Clutton-Brock T, Cooper G, Dawson A, Drife J, Garrod D, Harper A, Hulbert D, Lucas S, McClure J, Millward-Sadler H, Neilson J, Nelson-Piercy C, Norman J, O'Herlihy C, Oates M, Shakespeare J, de Swiet M, Williamson C, Beale V, Knight M, Lennox C, Miller A, Parmar D, Rogers J, Springett A. Saving Mothers' Lives: Reviewing maternal deaths to make motherhood safer: 2006-2008. The Eighth Report of the Confidential Enquiries into Maternal Deaths in the United Kingdom. BJOG. 2011 Mar;118(Suppl 1):1-203. doi: 10.1111/j.1471-0528.2010.02847.x. PMID 21356004
- [Background] Dall'Asta A, D'Antonio F, Saccone G, Buca D, Mastantuoni E, Liberati M, Flacco ME, Frusca T, Ghi T. Cardiovascular events following pregnancy complicated by pre-eclampsia with emphasis on comparison between early- and late-onset forms: systematic review and meta-analysis. Ultrasound Obstet Gynecol. 2021 May;57(5):698-709. doi: 10.1002/uog.22107. PMID 32484256
- [Background] Roberts LM, Davis GK, Homer CS. Pregnancy with gestational hypertension or preeclampsia: A qualitative exploration of women's experiences. Midwifery. 2017 Mar;46:17-23. doi: 10.1016/j.midw.2017.01.004. Epub 2017 Jan 10. PMID 28110162
- [Background] Bergink V, Laursen TM, Johannsen BM, Kushner SA, Meltzer-Brody S, Munk-Olsen T. Pre-eclampsia and first-onset postpartum psychiatric episodes: a Danish population-based cohort study. Psychol Med. 2015 Dec;45(16):3481-9. doi: 10.1017/S0033291715001385. Epub 2015 Aug 5. PMID 26243040
- [Background] Chesley LC, Cooper DW. Genetics of hypertension in pregnancy: possible single gene control of pre-eclampsia and eclampsia in the descendants of eclamptic women. Br J Obstet Gynaecol. 1986 Sep;93(9):898-908. doi: 10.1111/j.1471-0528.1986.tb08006.x. PMID 3768285
- [Background] Skjaerven R, Vatten LJ, Wilcox AJ, Ronning T, Irgens LM, Lie RT. Recurrence of pre-eclampsia across generations: exploring fetal and maternal genetic components in a population based cohort. BMJ. 2005 Oct 15;331(7521):877. doi: 10.1136/bmj.38555.462685.8F. Epub 2005 Sep 16. PMID 16169871
- [Background] Williams PJ, Broughton Pipkin F. The genetics of pre-eclampsia and other hypertensive disorders of pregnancy. Best Pract Res Clin Obstet Gynaecol. 2011 Aug;25(4):405-17. doi: 10.1016/j.bpobgyn.2011.02.007. Epub 2011 Mar 22. PMID 21429808
- [Background] Valenzuela FJ, Perez-Sepulveda A, Torres MJ, Correa P, Repetto GM, Illanes SE. Pathogenesis of preeclampsia: the genetic component. J Pregnancy. 2012;2012:632732. doi: 10.1155/2012/632732. Epub 2011 Dec 1. PMID 22175024
- [Background] Gallo DM, Wright D, Casanova C, Campanero M, Nicolaides KH. Competing risks model in screening for preeclampsia by maternal factors and biomarkers at 19-24 weeks' gestation. Am J Obstet Gynecol. 2016 May;214(5):619.e1-619.e17. doi: 10.1016/j.ajog.2015.11.016. Epub 2015 Nov 25. PMID 26627730
- [Background] Rolnik DL, Wright D, Poon LC, O'Gorman N, Syngelaki A, de Paco Matallana C, Akolekar R, Cicero S, Janga D, Singh M, Molina FS, Persico N, Jani JC, Plasencia W, Papaioannou G, Tenenbaum-Gavish K, Meiri H, Gizurarson S, Maclagan K, Nicolaides KH. Aspirin versus Placebo in Pregnancies at High Risk for Preterm Preeclampsia. N Engl J Med. 2017 Aug 17;377(7):613-622. doi: 10.1056/NEJMoa1704559. Epub 2017 Jun 28. PMID 28657417
- [Background] Rodriguez-Calvo J, Villalain C, Gomez-Arriaga PI, Quezada MS, Herraiz I, Galindo A. Prediction of perinatal survival in early-onset fetal growth restriction: role of placental growth factor. Ultrasound Obstet Gynecol. 2023 Feb;61(2):181-190. doi: 10.1002/uog.26116. PMID 36370447
- [Background] Crovetto F, Triunfo S, Crispi F, Rodriguez-Sureda V, Roma E, Dominguez C, Gratacos E, Figueras F. First-trimester screening with specific algorithms for early- and late-onset fetal growth restriction. Ultrasound Obstet Gynecol. 2016 Sep;48(3):340-8. doi: 10.1002/uog.15879. PMID 26846589
- [Background] Andrietti S, Silva M, Wright A, Wright D, Nicolaides KH. Competing-risks model in screening for pre-eclampsia by maternal factors and biomarkers at 35-37 weeks' gestation. Ultrasound Obstet Gynecol. 2016 Jul;48(1):72-9. doi: 10.1002/uog.15812. Epub 2016 May 30. PMID 26566592
- [Background] Ciobanu A, Wright A, Panaitescu A, Syngelaki A, Wright D, Nicolaides KH. Prediction of imminent preeclampsia at 35-37 weeks gestation. Am J Obstet Gynecol. 2019 Jun;220(6):584.e1-584.e11. doi: 10.1016/j.ajog.2019.01.235. Epub 2019 Feb 7. PMID 30738886
- [Background] Llurba E, Crispi F, Verlohren S. Update on the pathophysiological implications and clinical role of angiogenic factors in pregnancy. Fetal Diagn Ther. 2015;37(2):81-92. doi: 10.1159/000368605. Epub 2015 Feb 3. PMID 25659427
- [Background] Velez MP, Hamel C, Hutton B, Gaudet L, Walker M, Thuku M, Cobey KD, Pratt M, Skidmore B, Smith GN. Care plans for women pregnant using assisted reproductive technologies: a systematic review. Reprod Health. 2019 Jan 29;16(1):9. doi: 10.1186/s12978-019-0667-z. PMID 30696452
- [Background] Bhide A, Acharya G, Bilardo CM, Brezinka C, Cafici D, Hernandez-Andrade E, Kalache K, Kingdom J, Kiserud T, Lee W, Lees C, Leung KY, Malinger G, Mari G, Prefumo F, Sepulveda W, Trudinger B. ISUOG practice guidelines: use of Doppler ultrasonography in obstetrics. Ultrasound Obstet Gynecol. 2013 Feb;41(2):233-39. doi: 10.1002/uog.12371. No abstract available. PMID 23371348
- [Background] Lucas-Carrasco R. Reliability and validity of the Spanish version of the World Health Organization-Five Well-Being Index in elderly. Psychiatry Clin Neurosci. 2012 Oct;66(6):508-13. doi: 10.1111/j.1440-1819.2012.02387.x. PMID 23066768
- [Background] Pena-Chilet M, Roldan G, Perez-Florido J, Ortuno FM, Carmona R, Aquino V, Lopez-Lopez D, Loucera C, Fernandez-Rueda JL, Gallego A, Garcia-Garcia F, Gonzalez-Neira A, Pita G, Nunez-Torres R, Santoyo-Lopez J, Ayuso C, Minguez P, Avila-Fernandez A, Corton M, Moreno-Pelayo MA, Morin M, Gallego-Martinez A, Lopez-Escamez JA, Borrego S, Antinolo G, Amigo J, Salgado-Garrido J, Pasalodos-Sanchez S, Morte B; Spanish Exome Crowdsourcing Consortium; Carracedo A, Alonso A, Dopazo J. CSVS, a crowdsourcing database of the Spanish population genetic variability. Nucleic Acids Res. 2021 Jan 8;49(D1):D1130-D1137. doi: 10.1093/nar/gkaa794. PMID 32990755
- [Background] Plagnol V, Curtis J, Epstein M, Mok KY, Stebbings E, Grigoriadou S, Wood NW, Hambleton S, Burns SO, Thrasher AJ, Kumararatne D, Doffinger R, Nejentsev S. A robust model for read count data in exome sequencing experiments and implications for copy number variant calling. Bioinformatics. 2012 Nov 1;28(21):2747-54. doi: 10.1093/bioinformatics/bts526. Epub 2012 Aug 31. PMID 22942019